CLINICAL TRIAL: NCT06600009
Title: Treatment Persistence of Biologics in Patients with PsA in Japan; Retrospective Cohort Study Using a Claims Database (The FLYWAY Study)
Brief Title: Treatment Persistence of Biologics in Patients with PsA in Japan; Retrospective Cohort Study Using a Claims Database
Acronym: FLYWAY
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CAIN457FJP01
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Psoriatic Arthritis
Keywords: PSA
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab; Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Secukinumab: Patients had received secukinumab treatment.
  Interventions: Drug: Secukinumab
- Adalimumab: Patients had received adalimumab treatment.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Secukinumab — Patients had received secukinumab per their dosing regimens prior to this observational study.
  Groups: Secukinumab
Drug: Adalimumab — Patients had received adalimumab per their dosing regimens prior to this observational study.
  Groups: Adalimumab

SUMMARY:
This study was a retrospective non-interventional cohort study with secondary use of data from the Medical Data Vision (MDV) hospital-based database. The study setting was defined as follows:

* The inclusion period covered 01 February 2015 to 30 September 2020.
* The study period covered 01 August 2014 to 30 September 2021 inclusive.
* The index date was defined as the date of the first prescription of secukinumab or adalimumab within the inclusion period.
* The pre-index period was defined as the 6-month period before the index date (exclusive).
* Patients were followed until death, discontinuation of treatments of interest or end of the study period, whichever occurred first.

ELIGIBILITY:
Inclusion criteria:

* Having at least one biologic agent prescription of interest (secukinumab or adalimumab - princeps or biosimilars) recorded, in accordance with package insert, during the inclusion period (first prescription: index date).
* Having a confirmed diagnosis of PsA (the international classification of diseases, 10th revision [ICD-10]: L405) (at least 1 inpatient or outpatient claim without any doubtful flag) recorded during the pre-index period or at the index date.
* Being age 18 years or older at the index date.
* Having at least a 6-month pre-index period.

Bio-naive subgroup:

• Patients were considered as bio-naive if no record of any biologic agent prescriptions indicated for psoriasis or PsA (infliximab, adalimumab, certolizumab pegol, ustekinumab, risankizumab, guselkumab, secukinumab, ixekizumab, brodalumab - princeps or biosimilars) were retrieved during the pre-index period.

Exclusion Criteria:

* Having a biologic agent overdose (over 300 mg for secukinumab and over 80 mg for adalimumab) observed during the study period (off-label),
* Having at least one record of secukinumab (for secukinumab patients) or adalimumab (for adalimumab patients) retrieved during the pre-index period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Persistence of Secukinumab Treatment at One Year | 1 year

SECONDARY OUTCOMES:
Sex | Baseline
Age | Baseline
Number of Patients, Categorized by Medical Facility Department | Baseline
Height | Baseline
Weight | Baseline
Body Mass Index (BMI) | Baseline
Time from PsA Diagnosis to Index Date, Categorized by Medical Facility Department | Up approximately 6 months
Number of Patients with Comorbidities, by Category | Baseline
Number of Patients on Concomitant Treatments | Baseline
C-reactive Protein (CRP) | Baseline
Change in C-reactive Protein (CRP) Since Administration of Secukinumab or Adalimumab in Patients Still Treated with the Drug at the End of Follow-up | Up to approximately 5 years
Change in C-reactive Protein (CRP) Since Administration of Secukinumab or Adalimumab in Patients Who Discontinued the Drug | Up to approximately 5 years
Time from Index Date to the Start of Methotrexate Add-on | Up to approximately 5 years
Time from Index Date to Methotrexate Discontinuation in Methotrexate Naive Patients at Index Date | Up to approximately 5 years
Time from Index Date to Methotrexate Discontinuation in Methotrexate Experienced Patients at Index Date | Up to approximately 5 years
Secukinumab/adalimumab Dose at the Start of Methotrexate Add-on | Up to approximately 5 years
Secukinumab/adalimumab Dose at Methotrexate Discontinuation | Up to approximately 5 years
Number of Patients with Methotrexate Add-on During Follow-up | Up to approximately 5 years
Average Secukinumab/adalimumab Dose at Index Date | Baseline
Number of Patients with Persistence of Secukinumab or Adalimumab Treatment | 24 weeks, 1 year, 1.5 years, 2 years, 2.5 years, and 3 years
Time from PsA Diagnosis to Index Date for Adalimumab Patients | Up approximately 6 months
Number of Adalimumab Patients, Categorized by Medical Facility | Baseline
Number of Patients with Presence or Absence of Methotrexate | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharma K.K., Tokyo, Japan